CLINICAL TRIAL: NCT07031219
Title: Syndemic Triple HIV/HBV/HCV Virus Screening Via EMR Automation at Primary Care Clinics
Brief Title: HIV/HBV/HCV Triple Screening in Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Mamta K. Jain, MD,MPH, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU20240019; IN-US-973-7442 (Other Grant/Funding Number: Gilead)
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: HIV; HBV (Hepatitis B Virus); HCV
Keywords: screening; provider orders; quality improvement
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: This is a within-subjects repeated-measures unblinded design. All providers (participants) will have encounters randomized to control (no alert) or intervention (alert) throughout the duration of the study. Therefore, all providers (participants) are technically assigned to the same "study arm".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Randomized encounters (Other): For participating providers, each of their encounters will be randomized to either control (no alert; no changes to EMR interface; standard of care) or intervention (alert linked to triple testing orders will trigger when the provider attempts to order a screening test for HIV, hepatitis B, or hepatitis C). Since randomization will occur at the encounter level, participating providers will randomly experience control and intervention encounters throughout the duration of the study.
  Interventions: Other: electronic medical record alert linked to orders

INTERVENTIONS:
Other: electronic medical record alert linked to orders — An electronic medical record alert linked to triple testing orders will be built specifically for this study. An order for a screening blood test for any of the three bloodborne viruses (BBVs; i.e. HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV)) will trigger an electronic medical record alert linked to orders for screening blood tests for all three BBVs to be selected by default. If participants accept the alert, the individual BBV order that triggered the alert will be replaced with the pre-selected screening orders for all three BBVs. If the participants dismiss the alert, the individual BBV screening test order that triggered the alert will be accepted without the addition of screening test orders for the other two BBVs. This alert with linked orders will only be available to participating providers throughout the duration of the study, and will only activate for encounters randomized to "intervention" encounters.

SUMMARY:
Design:

This will be a within-subjects repeated-measures design, testing an electronic medical record pop-up alert linked to order panels for screening blood tests for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV). Study participants will be primary care providers. For each participating provider, their encounter will be randomized to either control (no alert; no changes to EMR interface) or an alert with triple-testing order panel intervention arm (alert linked to order panel with screening tests for all three bloodborne viruses (BBVs) selected by default; the alert will be triggered when a provider attempts to order a screening test for at least one BBV). The alert linked to triple testing orders will only be triggered if the provider orders a virus BBV screening test based on their normal practice and standard of care for their patient. Providers will see which orders are selected prior to signing (finalizing) them; therefore, this study will be unblinded. To mitigate the effect of unblinding, randomization will occur at the encounter level which will lead to providers experiencing both the control and intervention conditions randomly throughout the duration of the study.

Outcomes/endpoints:

The investigators will compare incidences of HIV, HBV, and HCV diagnoses between the two encounter conditions, estimate number of cases missed by not triple-testing, estimate laboratory costs per condition, and measure patient encounters per condition.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient primary care adult providers at participating institutions
* Providers who provide consent to participate in this study.
* Providers must intend to continue their current practice for at least 12 months.
* Providers with at least 12 months experience in their current practice.

Exclusion Criteria:

* Providers who do not consent to participate
* Sub-specialty providers
* Pediatric providers
* Providers who anticipate leaving their current practice within the next 12 months (i.e. providers who plan to retire, move, etc.).
* Providers with less than 12 months experience in their current practice (i.e. new providers or trainees who joined the practice within the last year)
* Note: family medicine and med/peds providers can participate, but only for their adult patients. The intervention alert+order panel and any data collection will be restricted to adult patients ≥ 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Bloodborne virus (BBV) screening tests | 24 months total: from 12 months pre-enrollment through the end of study participation (i.e. maximum of 1 year of participation)
  For total bloodborne virus (BBV) screening tests (HIV, hepatitis B virus (HBV), and hepatitis C virus (HCV) combined) and each individual BBV (HIV, HBV, or HCV independently), the investigators will measure the number of screening tests: 1) ordered, 2) performed, 3) with a positive result, 4) with a negative result: overall across all encounters, and compared between control and intervention encounters as well as normalized to the providers' pre-study baseline

SECONDARY OUTCOMES:
Prevalences of bloodborne viruses (BBVs) | 24 months total: from 12 months pre-enrollment through the end of study participation (i.e. maximum of 1 year of participation)
  Prevalences of HIV, hepatitis B virus (HBV), and hepatitis C virus (HCV) as well as BBV co-infections among patients of participating providers overall across all encounters, and compared between control and intervention encounters as well as normalized to the providers' pre-study baseline
Incidences of bloodborne viruses (BBVs) | 24 months total: from 12 months pre-enrollment through the end of study participation (i.e. maximum of 1 year of participation)
  Incidences of HIV, hepatitis B virus (HBV), and hepatitis C virus (HCV) as well as BBV co-infections among patients of participating providers overall across all encounters, and compared between control and intervention encounters as well as normalized to the providers' pre-study baseline
Number of patient encounters required to make a virus diagnosis and link patients to care | 24 months total: from 12 months pre-enrollment through the end of study participation (i.e. maximum of 1 year of participation)
  Number of patient encounters required to make a virus diagnosis and link patients to care overall across all encounters, and compared between control and intervention encounters as well as normalized to the providers' pre-study baseline
Cost efficiency analysis | 24 months total: from 12 months pre-enrollment through the end of study participation (i.e. maximum of 1 year of participation)
  Assess and determine cost efficiency via analysis of laboratory costs by estimating laboratory costs per patient and per new diagnosis overall across all encounters, and compared between control and intervention encounters as well as normalized to the providers' pre-study baseline
Repeated BBV tests | 24 months total: from 12 months pre-enrollment through the end of study participation (i.e. maximum of 1 year of participation)
  Measure frequencies of repeated tests before and after excluding those with a known BBV diagnosis prior to the study across all encounters, and compared between control and intervention encounters as well as normalized to the providers' pre-study baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mamta K Jain, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No